CLINICAL TRIAL: NCT04004754
Title: Documenting Clinical Outcomes of Patients Receiving Miltefosine for the Treatment of Complicated Cutaneous Leishmaniasis in Ethiopia
Brief Title: Outcomes of Complicated CL in Ethiopia Treated With Miltefosine
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: University of Gondar (Other); Boru Meda Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1243/18
Record Dates: First submitted 2019-06-26; First posted 2019-07-02 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Cutaneous Leishmaniases
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — miltefosine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Routinely collected skin slit smears from the lesions were stored. Scrapings of these skin slit smears were analyzed by PCR and a selected group will be analyzed for species typing.
  Patients could opt out of biospecimen storage and use for study purposes.
Oversight: FDA-regulated Device: No

GROUPS / COHORTS (2):
- Complicated CL in Gondar: Patients treated with miltefosine in Gondar will be followed up to see outcomes of treatment
  Interventions: Drug: Miltefosine (administration is not part of study procedures)
- Complicated CL in Boru Meda: Patients treated with miltefosine in Boru Meda hospital will be followed up to see outcomes of treatment
  Interventions: Drug: Miltefosine (administration is not part of study procedures)

INTERVENTIONS:
Drug: Miltefosine (administration is not part of study procedures) — Patients who receive miltefosine in the routine setting will be asked to participate in the study to document their outcomes

SUMMARY:
Cutaneous Leishmaniasis in Ethiopia causes severe dermatological mutilations. Forms that require systemic treatment are cLCL, MCL, and DCL. National guidelines recommend equally all drugs that are also used for VL treatment. Miltefosine is one of these recommended medications but remains underused due to scarcity of drugs.

Outcomes of patients receiving miltefosine have never been documented systematically in Ethiopia until today. This is needed to provide evidence to advocate for increased access to miltefosine in Ethiopia, and to establish baseline data for future research on CL treatment options. The aim of this study is to document treatment outcomes of patients with cLCL, MCL, and DCL receiving systemic treatment using miltefosine within a routine care setting located in an endemic area in Ethiopia.

ELIGIBILITY:
Inclusion Criteria:

* Parasitologically or clinically confirmed diagnosis of Leishmaniasis
* Clinical routine care decision to initiate miltefosine

Exclusion Criteria:

* Medical emergencies, underlying chronic conditions, or other circumstances that make participation in this study medically or otherwise inadvisable

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with complicated CL receiving miltefosine
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-06-11 (Actual)

PRIMARY OUTCOMES:
Assess final treatment response | Day 90
  proportion of index lesions with cure, good, partial and no treatment response

SECONDARY OUTCOMES:
Early and late treatment response | Day 28, Day 180
  Proportion of index lesions with cure, good, partial and no treatment response at Day 28 and Day 180
Treatment failure | Day 90, Day 180
  Proportion of index lesions with relapse or failure at Day 90 and Day 180
Adherence | Day 28
  Proportion of patients with excellent (0 missed), good (1-3 missed), mediocre (4-8 missed), and poor (<=9 missed) adherence
Predictors of cure | Day 90
  Covariate-adjusted risk ratios of factors associated with cure of index lesions at Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Johan van Griensven, MD,PhD, Study Director — Institute of Tropical Medicine
Locations (2):
- Ethiopia (2):
  - Boru Meda Hospital, Boru
  - Gondar University Hospital, Gonder

IPD SHARING:
Plan to Share IPD: Yes
Data can be made available to research by means of a managed access procedure
Supporting Information: Study Protocol
Time Frame: After completion of the primary publication
Access Criteria: Managed access procedure - applicants need to fill out a data access request form
URL: https://www.itg.be/E/data-sharing-open-access

REFERENCES:
- [Derived] van Henten S, Tesfaye AB, Abdela SG, Tilahun F, Fikre H, Buyze J, Kassa M, Cnops L, Pareyn M, Mohammed R, Vogt F, Diro E, van Griensven J. Miltefosine for the treatment of cutaneous leishmaniasis-A pilot study from Ethiopia. PLoS Negl Trop Dis. 2021 May 28;15(5):e0009460. doi: 10.1371/journal.pntd.0009460. eCollection 2021 May. PMID 34048461